CLINICAL TRIAL: NCT03802448
Title: Effect of Myofascial Release on Electrophysiological and Clinical Measures of Pregnant Women With Carpal Tunnel Syndrome
Brief Title: Myofascial Release on Electrophysiological Measures of Pregnant Women With CTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HAhmed, Deputy Director of Quality Assurance Unit, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/011/001990
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2013-05

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): composed of fifteen pregnant women who only wore a natural wrist splint during sleeping for 4 weeks.
  A neutral wrist splint was worn by all pregnant women in both groups daily at night, only all through the study time (4 weeks). This neutral wrist splint was used to keep the wrist in a straight position (neutral position) and to prevent the extreme wrist motion (flexion and extension) while sleeping
  Interventions: Device: Control group
- Study group (Experimental): a myofascial release in addition to wearing a natural wrist splint during sleeping for 4 weeks.
  Myofascial wrist retinaculum (Transverse carpal ligament) release.
  • Second part; Interosseous membrane and forearm muscles myofascial release (Bilateral thumb pressure technique).
  Interventions: Combination Product: Study group; Device: Control group

INTERVENTIONS:
Combination Product: Study group — Each pregnant woman in the study group received myofascial release technique, 3 sessions/week for 4 weeks. a myofascial release in addition to wearing a natural wrist splint during sleeping for 4 weeks.
  Myofascial wrist retinaculum (Transverse carpal ligament) release.
  • Second part; Interosseous membrane and forearm muscles myofascial release (Bilateral thumb pressure technique).
  Arms: Study group
Device: Control group — A neutral wrist splint was worn by all pregnant women in both groups daily at night, only all through the study time (4 weeks). This neutral wrist splint was used to keep the wrist in a straight position (neutral position) and to prevent the extreme wrist motion (flexion and extension) while sleeping.

SUMMARY:
Objective: To explore the effect of myofascial release on electrophysiological and clinical measures of pregnant women with carpal tunnel syndrome (CTS).

Design: Randomized controlled trial. Methods: Thirty pregnant women had CTS, their age ranged from 25-35 years, were randomized into two equal groups. The control group only wore a natural wrist splint during sleeping for 4 weeks, while the study group received a myofascial release in addition to wearing a natural wrist splint during sleeping for 4 weeks. All pregnant women in both groups were evaluated pre and post-treatment through median nerve distal motor latency (DML) and Boston carpal tunnel questionnaire (BCTQ) to assess pain, numbness & tingling sensation severity and hand function.

DETAILED DESCRIPTION:
Design This study was designed as a prospective, randomized, controlled trial. The Research Ethical Committee of the Faculty of Physical Therapy, Cairo University approved this study. The study was conducted between May 2013 and April 2014.

Participants A sample of thirty pregnant women were recruited from the Obstetric Out-patient Clinic, El-Sahel Teaching Hospital, Cairo, Egypt. To be included in the study, the participants were chosen pregnant women at early of the third trimester complaining from idiopathic CTS (pain, numbness and tingling of the hand), which was confirmed by electrophysiological examination (i.e. delayed median DML < 3.9 msec) as well as positive Phalen's test. Pregnant women having bilateral and unilateral CTS affection participated but the dominant hand data only were enrolled in this study. Their ages ranged from 25 to 35 years old, their body mass index (BMI) did not exceed 34 Kg/m2 and their gravidity number ranged from 1 to 3 times. The participants were excluded if they had other predisposing causes for CTS and/or neuromuscular diseases that might affect median nerve transmission such as diabetes mellitus, pre-eclampsia, rheumatoid arthritis, previous CTS symptoms, acute hand trauma, cervical spondylosis, previous surgeries in the forearm involving the median nerve, peripheral neuropathy and pronator teres syndrome. All pregnant women did not receive any physical or medical therapy for treating CTS complains and had no serious medical problems as pacemaker and heart diseases that might interfere with electrophysiological testing.

Randomization Informed consent was signed by each participant after explaining the nature, purpose, and benefits of the study, informing them of their right to refuse or withdraw at any time, and about the confidentiality of any obtained data. The pregnant women were randomly assigned into two equal groups (control group and study group), a computer-based randomization program. No dropping out of subjects from the study after randomization.

Interventions Participants were randomly assigned into; Control group composed of fifteen pregnant women who only wore a natural wrist splint during sleeping for 4 weeks. Study group composed of fifteen pregnant women who received a myofascial release in addition to wearing a natural wrist splint during sleeping for 4 weeks.

Neutral wrist splint A neutral wrist splint was worn by all pregnant women in both groups daily at night, only all through the study time (4 weeks). This neutral wrist splint was used to keep the wrist in a straight position (neutral position) and to prevent the extreme wrist motion (flexion and extension) while sleeping.

Myofascial release technique

Each pregnant woman in the study group received myofascial release technique, 3 sessions/week for 4 weeks. The position of treatment was long sitting with the back fully supported, the dominant palm and forearm exposed and rested comfortably. Myofascial release technique was divided into two parts:

* First part; Myofascial wrist retinaculum (Transverse carpal ligament) release: The physical therapist placed her fourth and fifth fingers of both hands between the pregnant woman's fourth and fifth fingers and first and second fingers of the palmar surface and extension of the pregnant woman's wrist was introduced. The Physical therapist's thumbs overlie the lateral and medial attachments of the wrist flexor retinaculum and transverse distraction to the retinaculum was applied until relaxation of the soft tissue or release of the restriction was achieved (for about 30 seconds) then relaxation time was about 10 seconds. 15 repetitions were made in each session, three sessions per week for four weeks.
* Second part; Interosseous membrane and forearm muscles myofascial release (Bilateral thumb pressure technique): Gentle force was applied ventrally on the forearm through 2 hands grasping the pregnant woman's distal forearm with the thumbs contacting the anterior aspect of the forearm muscles and interosseous membrane while the index fingers grasping the posterior aspect of the forearm to engage the soft tissues cephalad until a barrier of tissue motion was reached and hold for about 30 seconds then relaxation time was about 10 seconds. 15 repetitions were made in each session, three sessions per week for four weeks Outcome Measures

Median nerve DML:

It was done for all the pregnant women in both groups before participation in this study to confirm their diagnosis of CTS and also after the end of the treatment.

Each pregnant woman in both groups was asked to evacuate her bladder to be more relaxed and then she was informed about the aim and steps of the test while she was seated on a wooden chair and her back was supported. The dominant forearm was in supinated position, rested on the examining table and the elbow joint held slightly flexed. The pregnant woman's body temperature was measured with an oral mercury thermometer and if it was normal, the test procedure was carried out and also the room temperature was adjusted at 22 °C, which controlled by an air conditioner as median nerve DML could be affected by the pregnant woman temperature as well as the room temperature.

Before electrode placement, the areas used for recording, stimulating or ground points were cleaned by alcohol to clean the skin to decrease its resistance. Further reduction of impedance was obtained by using conducting gel on the surface of the recording electrodes.

Then, the electromyography was calibrated and the parameters of the apparatus were adjusted as follows: Time base at 5.0 milliseconds/division, the sensitivity at 4000.0 volts/division and the intensity according to the site of stimulation; it was about 7 mA at the wrist stimulation and 12 mA for the elbow stimulation [7].

After the end of the previous preparation, the active recording electrode was placed on the motor point of the abductor pollicis brevis muscle and the reference recording electrode on the tip of the thumb. They were fixed to the hand by adhesive plaster straps. The bipolar stimulating electrode was placed above the wrist joint between the tendons of palmaris longus and the flexor carpi radialis muscles on the course of the median nerve, with the negative pole distal toward the active recording electrode, and the positive pole proximal to stimulate the median nerve. The ground electrode was placed on the distal wrist crease midway between the stimulating and recording electrodes, 7 mA was used at wrist stimulation.

Then, the bipolar stimulating electrode was placed in the cubital fossa, just medial to the biceps tendon, with the negative pole distal toward the active recording electrode, and the positive pole proximal. The recording electrodes were applied at the same locations as in recording at wrist level. 12 mA was used at elbow stimulation.

BCTQ:

It was self-applied and evaluated the severity of symptoms and the functional status of patients with CTS. It had comprehensive framework, good validity, reliability and responsiveness in the hands of the researchers [8]. The questionnaire compromised two scales, a symptoms severity scale (SSS) and a functional status scale (FSS). The SSS evaluated symptoms regarding severity, frequency and time. The FSS evaluated how the syndrome affects daily life. Questions concerning SSS composed of 11 questions addressing: Pain intensity during day time and night time, time of pain during the day, dormancy, weakness, tingling sensation at night, frequency of that night tingling sensation and skill. Each question had five answers numbered from 0 point (no symptoms) to 4 points (most severe). Questions concerning FSS consisted of daily activities that were performed by most individuals and were commonly affected by CTS. The patients rated their ability to perform the activity on a scale that ranged from 1 point (no difficulty with the activity) to 5 points (cannot perform the activity at all). The overall score for the FSS was the mean of the ratings on the daily activities. This questionnaire was performed before and after treatment for both groups.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the study, the participants were chosen pregnant women at early of the third trimester complaining from idiopathic CTS (pain, numbness and tingling of the hand), which was confirmed by electrophysiological examination (i.e. delayed median DML < 3.9 msec) as well as positive Phalen's test. Pregnant women having bilateral and unilateral CTS affection participated but the dominant hand data only were enrolled in this study. Their ages ranged from 25 to 35 years old, their body mass index (BMI) did not exceed 34 Kg/m2 and their gravidity number ranged from 1 to 3 times.

Exclusion Criteria:

* The participants were excluded if they had other predisposing causes for CTS and/or neuromuscular diseases that might affect median nerve transmission such as diabetes mellitus, pre-eclampsia, rheumatoid arthritis, previous CTS symptoms, acute hand trauma, cervical spondylosis, previous surgeries in the forearm involving the median nerve, peripheral neuropathy and pronator teres syndrome. All pregnant women did not receive any physical or medical therapy for treating CTS complains and had no serious medical problems as pacemaker and heart diseases that might interfere with electrophysiological testing

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
change of Median nerve Distal Motor Latency | pretreatment, after 4 weeks of the treatment
  , the active recording electrode was placed on the motor point of the abductor pollicis brevis muscle and the reference recording electrode on the tip of the thumb. They were fixed to the hand by adhesive plaster straps. The bipolar stimulating electrode was placed above the wrist joint between the tendons of palmaris longus and the flexor carpi radialis muscles on the course of the median nerve, with the negative pole distal toward the active recording electrode, and the positive pole proximal to stimulate the median nerve. The ground electrode was placed on the distal wrist crease midway between the stimulating and recording electrodes, 7 mA was used at wrist stimulation

SECONDARY OUTCOMES:
change of Boston carpal tunnel questionnaire (BCTQ) | pretreatment, after 4 weeks of the treatment
  The questionnaire compromised two scales, a symptoms severity scale (SSS) and a functional status scale (FSS)

IPD SHARING:
Plan to Share IPD: Undecided